CLINICAL TRIAL: NCT02658214
Title: A Phase Ib Study to Evaluate the Safety and Tolerability of Durvalumab and Tremelimumab in Combination With First-Line Chemotherapy in Patients With Advanced Solid Tumors.
Brief Title: Durvalumab and Tremelimumab in Combination With First-Line Chemotherapy in Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D419SC00001
Record Dates: First submitted 2016-01-11; First posted 2016-01-18 (Estimated); Last update posted 2020-08-20 (Actual); Status verified 2020-08

CONDITIONS: Small Cell Lung Carcinoma; Carcinoma, Squamous Cell of Head and Neck; Stomach Neoplasms; Triple Negative Breast Neoplasms; Ovarian Neoplasms; Fallopian Tube Neoplasms; Peritoneal Neoplasms; Esophagogastric Junction Neoplasms; Carcinoma, Pancreatic Ductal; Esophageal Squamous Cell Carcinoma
Keywords: durvalumab, tremelimumab, metastatic, solid tumors, immuno-oncology, first-line chemotherapy, esophageal, pancreatic
MeSH Terms: conditions — Small Cell Lung Carcinoma; Squamous Cell Carcinoma of Head and Neck; Stomach Neoplasms; Triple Negative Breast Neoplasms; Ovarian Neoplasms; Fallopian Tube Neoplasms; Peritoneal Neoplasms; Carcinoma, Pancreatic Ductal; Esophageal Squamous Cell Carcinoma; Neoplasm Metastasis | interventions — CP protocol; EC regimen; Gemcitabine; Carboplatin; 130-nm albumin-bound paclitaxel; Oxaliplatin; Fluorouracil; Leucovorin; durvalumab; tremelimumab; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Cohort 1 (Experimental): ovarian/peritoneal/fallopian tube cancer and squamous cell carcinoma of the head and neck (SCCHN)
  Interventions: Drug: paclitaxel + carboplatin; Biological: durvalumab; Biological: tremelimumab
- Cohort 2 (Experimental): Small-cell lung cancer (SCLC)
  Interventions: Drug: carboplatin + etoposide; Biological: durvalumab; Biological: tremelimumab
- Cohort 3 (Experimental): Triple-negative breast cancer (TNBC)
  Interventions: Drug: gemcitabine + carboplatin; Biological: durvalumab; Biological: tremelimumab
- Cohort 4 (Experimental): Triple-negative breast cancer (TNBC)
  Interventions: Drug: nab-paclitaxel (paclitaxel-albumin) + carboplatin; Biological: durvalumab; Biological: tremelimumab
- Cohort 5 (Experimental): Gastric/gastro-esophageal junction (GEJ)
  Interventions: Drug: oxaliplatin + 5-fluorouracil (5FU) + leucovorin (calcium folinate/folinic acid); Biological: durvalumab; Biological: tremelimumab
- Cohort 6 (Experimental): Pancreatic ductal adenocarcinoma (PDAC)
  Interventions: Biological: durvalumab; Biological: tremelimumab; Drug: nab-paclitaxel (paclitaxel-albumin) + gemcitabine
- Cohort 7 (Experimental): Esophageal squamous cell carcinoma (ESCC)
  Interventions: Biological: durvalumab; Biological: tremelimumab; Drug: cisplatin + 5-fluorouracil (5FU)

INTERVENTIONS:
Drug: paclitaxel + carboplatin — IV infusion
  Other Names: Platinum based Standard of Care Chemotherapy
  Arms: Cohort 1
Drug: carboplatin + etoposide — IV infusion
  Other Names: Platinum based Standard of Care Chemotherapy
  Arms: Cohort 2
Drug: gemcitabine + carboplatin — IV infusion
  Other Names: Platinum based Standard of Care Chemotherapy
  Arms: Cohort 3
Drug: nab-paclitaxel (paclitaxel-albumin) + carboplatin — IV infusion
  Other Names: Platinum based Standard of Care Chemotherapy
  Arms: Cohort 4
Drug: oxaliplatin + 5-fluorouracil (5FU) + leucovorin (calcium folinate/folinic acid) — IV infusion and bolus administration
  Other Names: Platinum based Standard of Care Chemotherapy
  Arms: Cohort 5
Biological: durvalumab — IV infusion
  Other Names: MEDI4736
Biological: tremelimumab — IV infusion
Drug: nab-paclitaxel (paclitaxel-albumin) + gemcitabine — IV infusion
  Other Names: Standard of Care Chemotherapy
  Arms: Cohort 6
Drug: cisplatin + 5-fluorouracil (5FU) — IV infusion
  Other Names: Platinum based Standard of Care Chemotherapy
  Arms: Cohort 7

SUMMARY:
Durvalumab and Tremelimumab in combination with first-line chemotherapy in the following indications: Ovarian/peritoneal/fallopian tube cancer, SCCHN, TNBC, SCLC and gastric/GEJ cancer, PDAC, ESCC.

DETAILED DESCRIPTION:
7 cohorts of first-line chemotherapy regimens combined with durvalumab + tremelimumab.

This study will evaluate the safety and tolerability of durvalumab (MEDI4736) + tremelimumab in combination with first line chemotherapy regimens in patients with locally advanced or metastatic solid tumors: ovarian/peritoneal/fallopian tube cancer, squamous cell carcinoma of the head and neck (SCCHN), triple negative breast cancer (TNBC), small cell lung carcinoma (SCLC), and gastric/gastro-esophageal junction (GEJ) cancer, pancreatic ductal adenocarcinoma (PDAC) and esophageal squamous cell carcinoma (ESCC).

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years
2. Written informed consent
3. Patients with histologically or cytologically documented chemotherapy-naïve locally advanced unresectable or metastatic ovarian/peritoneal/fallopian tube cancer, SCCHN, TNBC, SCLC, gastric cancer/GEJ, PDAC and ESCC.
4. ECOG performance status of 0 or 1
5. Patients must be considered suitable candidates for, and able to receive, first line chemotherapy for metastatic disease
6. At least 1 lesion, not previously irradiated, that can be accurately measured at baseline
7. No prior exposure to immune-mediated therapy
8. Adequate organ and marrow function as defined below

Exclusion Criteria:

1. Receipt of any investigational anticancer therapy within 28 days or 5 halflives, whichever is longer, prior to the first dose of study treatment
2. Brain metastases or spinal cord compression unless asymptomatic or treated and stable off steroids and anti-convulsants for at least 1 month prior to study treatment
3. Any unresolved Grade ≥2 toxicity from previous anticancer therapy
4. Active or prior documented autoimmune or inflammatory disorders
5. Uncontrolled intercurrent illness, including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs from study drugs, or compromise the ability of the patient to give written informed consent
6. Mean QT interval corrected for heart rate using Fridericia's formula (QTcF) ≥470 ms 20. Active tuberculosis
7. Active infection including tuberculosis, hepatitis B, hepatitis C, or human immunodeficiency virus (HIV)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2016-04-28 (Actual); Primary Completion 2019-11-14 (Actual); Study Completion 2019-11-14 (Actual)

PRIMARY OUTCOMES:
Laboratory findings (including: clinical chemistry, hematology, and urinalysis) | Throughout the study, approximately three years
  To assess the safety and tolerability profile of first-line chemotherapy in combination with durvalumab + tremelimumab
Incidence of Adverse Events | Throughout the study, approximately three years
  To assess incidence of Adverse Events for the safety and tolerability profile of first-line chemotherapy in combination with durvalumab and tremelimumab
Tumor assessment based on RECIST 1.1 (for cohort 6 only) | Throughout the study, approximately three years (for cohort 6 only)
  To estimate the objective response rate (ORR) of durvalumab + tremelimumab + chemotherapy (for cohort 6 only)

CONTACTS AND LOCATIONS:
Locations (3):
- Japan (2):
  - Research Site, Chūōku
  - Research Site, Kashiwa
- Research Site, Seoul, South Korea

REFERENCES:
- [Derived] Lee DH, Kim HR, Keam B, Kato K, Kuboki Y, Gao H, Yovine A, Robbins SH, Ahn MJ. Safety and tolerability of first-line durvalumab with tremelimumab and chemotherapy in esophageal squamous cell carcinoma. Cancer Med. 2023 Aug;12(15):16066-16075. doi: 10.1002/cam4.6260. Epub 2023 Jul 25. PMID 37489066
- See also: Results of this clinical trial are available on www.astrazenecaclinicaltrials.com — https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Search